CLINICAL TRIAL: NCT00976001
Title: Open, Randomized Follow-up Pilot Study After a First Stroke
Brief Title: Follow-up Pilot Study After a First Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Lennart Welin, Department of Medicine, Lidkoeping Hospital, SE-531 85 Lidkoeping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VGSKAS-2300
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Stroke
Keywords: Follow-up after stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up at an out-patient stroke unit (Other): Information, measurement of handicap, further rehabilitation efforts, drug therapy for secondary prevention of stroke.
  Interventions: Other: Information, further rehabilitation, additional drugs to prevent recurrent stroke
- Follow-up with the general practitioner (Other)
  Interventions: Other: As the general practitioner wants to do

INTERVENTIONS:
Other: Information, further rehabilitation, additional drugs to prevent recurrent stroke
  Arms: Follow-up at an out-patient stroke unit
Other: As the general practitioner wants to do
  Arms: Follow-up with the general practitioner

SUMMARY:
This is a randomized follow-up study after discharge from a stroke unit after a first stroke. The patients are randomized either to follow-up at a special out-patient stroke unit or with their general practitioners. The hypothesis is that follow-up with specialists is superior to follow-up with general practitioners. Endpoints are mortality, recurrent stroke and handicap measured with different scales.

ELIGIBILITY:
Inclusion Criteria:

* first stroke (ischemic or hemorrhagic)
* age below 85 years
* living at home before the stroke

Exclusion Criteria:

* modified Rankin scale 5 points
* other severe disease
* expected survival less than one year
* severe dementia
* drug or alcohol abuse

Max Age: 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2003-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Total mortality | 3.5 years

SECONDARY OUTCOMES:
Recurrent stroke | 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke unit, Department of Medicine, Lidkoeping hospital, Lidköping, Sweden